CLINICAL TRIAL: NCT05408273
Title: Vitamin D Effects on Microvascular Function and Cardiovascular Risk Factors on Postmenopausal Women
Brief Title: Vitamin D and Microvascular Function in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, THAYSA FERNANDES LACERDA ROCHA COSTA, Principal Investigator on the Clinical and Experimental Pathophysiology Program, Rio de Janeiro State University
Other Study IDs: 31448514.1.0000.5282
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Menopause Related Conditions; Vitamin D Deficiency; Cardiovascular Diseases
Keywords: Menopause; Vitamin D; Microvascular Circulation; Laser Doppler Flowmetry
MeSH Terms: conditions — Vitamin D Deficiency; Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postmenopausal women: Associations of 25(OH)D to adiposity, blood pressure, fasting aldosterone, insulin, glucose and lipid profile, HOMA-IR, parathormone and microvascular function, assessed by laser-Doppler flowmetry at cutaneous site, were investigated.
  Interventions: Diagnostic Test: Blood samples and Microvascular function assessment evaluated through laser-Doppler flowmetry by the LASER speckle contrast analysis (LASCA) device

INTERVENTIONS:
Diagnostic Test: Blood samples and Microvascular function assessment evaluated through laser-Doppler flowmetry by the LASER speckle contrast analysis (LASCA) device — We enrolled 39 non-smokers, low CVR postmenopausal women, with less than 10 years of hypoestrogenism. Associations of 25(OH)D to adiposity, blood pressure, fasting aldosterone, insulin, glucose and lipid profile, HOMA-IR, parathormone and microvascular function, assessed by laser-Doppler flowmetry at cutaneous site, were investigated

SUMMARY:
Many observational studies have demonstrated links between serum levels of 25-hydroxyvitamin D [25(OH)D] and cardiovascular risk (CVR) factors. Microvascular dysfunction relates not only to CVR but also to metabolic disease. Since cardiovascular disease (CVD) is the leading cause of death in postmenopausal women, it would be relevant to confirm this relationship. Maybe further studies would show that the correction of hypovitaminosis D could minimize the CVR. Our objective with this clinical trail is to analyze if vitamin D status is related to microvascular function and conventional cardiovascular risk (CVR) factors in postmenopausal women. For that we enrolled, in a pilot cross-sectional study, 39 non-smokers, low CVR postmenopausal women, with less than 10 years of hypoestrogenism and associations of 25(OH)D to adiposity, blood pressure, fasting aldosterone, insulin, glucose and lipid profile, HOMA-IR, parathormone and microvascular function, assessed by laser-Doppler flowmetry at cutaneous site, were investigated.

ELIGIBILITY:
Inclusion Criteria:

Women between 45-60 years with clinical/laboratory criteria of menopause and duration of hypoestrogenism < 10 years. Menopause was spontaneous (at least one year of amenorrhea) or surgical (after bilateral oophorectomy). In hysterectomized women, ovarian failure was estimated by the history of vasomotor symptoms and serum levels of follicle-stimulating hormone (FSH) > 35 mU/mL and estradiol levels <20 pg/mL.

Exclusion Criteria:

Current smokers, body mass index (BMI) >35 kg/m², systolic BP >160 mmHg and or diastolic BP > 100 mmHg, total cholesterol >280 mg/dL, presence of T2D, renal dysfunction and or liver disease, clinical manifestations of coronary heart disease, and previous history of revascularization or cardiovascular event.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women from the gonad outpatient clinic of the Teaching Unit Endocrinology Department at Pedro Ernesto University Hospital/University of State of Rio de Janeiro, which integrates the state network of the Unified Health System, and volunteers who may be recruited from other HUPE Services or externally.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Vitamin D status and microvascular function | 1 day
  Vitamin D status and its relation to microvascular function and conventional cardiovascular risk (CVR) factors in postmenopausal women.

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosenberry R, Nelson MD. Reactive hyperemia: a review of methods, mechanisms, and considerations. Am J Physiol Regul Integr Comp Physiol. 2020 Mar 1;318(3):R605-R618. doi: 10.1152/ajpregu.00339.2019. Epub 2020 Feb 5. PMID 32022580
- [Background] Zhang QY, Jiang CM, Sun C, Tang TF, Jin B, Cao DW, He JS, Zhang M. Hypovitaminosis D is associated with endothelial dysfunction in patients with non-dialysis chronic kidney disease. J Nephrol. 2015 Aug;28(4):471-6. doi: 10.1007/s40620-014-0167-8. Epub 2014 Dec 17. PMID 25515034
- [Background] Equils O, Naiki Y, Shapiro AM, Michelsen K, Lu D, Adams J, Jordan S. 1,25-Dihydroxyvitamin D inhibits lipopolysaccharide-induced immune activation in human endothelial cells. Clin Exp Immunol. 2006 Jan;143(1):58-64. doi: 10.1111/j.1365-2249.2005.02961.x. PMID 16367934
- [Background] Brewer LC, Michos ED, Reis JP. Vitamin D in atherosclerosis, vascular disease, and endothelial function. Curr Drug Targets. 2011 Jan;12(1):54-60. doi: 10.2174/138945011793591617. PMID 20795937
- [Background] Napoli C, de Nigris F, Williams-Ignarro S, Pignalosa O, Sica V, Ignarro LJ. Nitric oxide and atherosclerosis: an update. Nitric Oxide. 2006 Dec;15(4):265-79. doi: 10.1016/j.niox.2006.03.011. Epub 2006 Apr 15. PMID 16684613
- [Background] Vinet A, Morrissey C, Perez-Martin A, Goncalves A, Raverdy C, Masson D, Gayrard S, Carrere M, Landrier JF, Amiot MJ. Effect of vitamin D supplementation on microvascular reactivity in obese adolescents: A randomized controlled trial. Nutr Metab Cardiovasc Dis. 2021 Jul 22;31(8):2474-2483. doi: 10.1016/j.numecd.2021.04.025. Epub 2021 May 10. PMID 34090775
- [Background] Andrukhova O, Slavic S, Zeitz U, Riesen SC, Heppelmann MS, Ambrisko TD, Markovic M, Kuebler WM, Erben RG. Vitamin D is a regulator of endothelial nitric oxide synthase and arterial stiffness in mice. Mol Endocrinol. 2014 Jan;28(1):53-64. doi: 10.1210/me.2013-1252. Epub 2013 Jan 1. PMID 24284821
- [Background] Codoner-Franch P, Tavarez-Alonso S, Simo-Jorda R, Laporta-Martin P, Carratala-Calvo A, Alonso-Iglesias E. Vitamin D status is linked to biomarkers of oxidative stress, inflammation, and endothelial activation in obese children. J Pediatr. 2012 Nov;161(5):848-54. doi: 10.1016/j.jpeds.2012.04.046. Epub 2012 Jun 5. PMID 22677566
- [Background] Kim DH, Meza CA, Clarke H, Kim JS, Hickner RC. Vitamin D and Endothelial Function. Nutrients. 2020 Feb 22;12(2):575. doi: 10.3390/nu12020575. PMID 32098418
- [Background] Schmitt EB, Nahas-Neto J, Bueloni-Dias F, Poloni PF, Orsatti CL, Petri Nahas EA. Vitamin D deficiency is associated with metabolic syndrome in postmenopausal women. Maturitas. 2018 Jan;107:97-102. doi: 10.1016/j.maturitas.2017.10.011. Epub 2017 Oct 18. PMID 29169589